CLINICAL TRIAL: NCT03703349
Title: Preoperative Oral Magnesium Versus Standard of Care to Prevent Postoperative Atrial Fibrillation Following Coronary Surgery (POMAF-CS): A Randomized Controlled Trial
Brief Title: Preoperative Oral Magnesium to Prevent Postoperative Atrial Fibrillation Following Coronary Surgery (POMAF-CS)
Acronym: POMAF-CS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, Samia Madi Jebara, Professor, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEHDF 850
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease; Surgery--Complications
Keywords: Coronary artery surgery; oral magnesium; atrial fibrillation; Randomized controlled trial
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — Magnesium Sulfate; Magnesium

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to the 2 groups of treatment by blocks of 8. The randomization list will be computer-generated, with no factors for stratification. To reduce predictability of the random sequence, blocking will be made unavailable to those who assign interventions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: treatment concealment will be managed by the central pharmacy of the hospital, which will dispense treatment according to the randomization plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative oral Magnesium (Experimental): Magnesium sulfate 8 tablets (8 x 0.4 g) per day, PO, for the 3 days preceding the surgical intervention
  Interventions: Drug: Magnesium Sulfate
- Control (Placebo Comparator): Placebo oral tablet, for Magnesium Sulfate tablets, PO, for the 3 days preceding the surgical intervention
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium sulfate will be prescribed by the surgeon / Anesthesiologist and will be taken orally by the patient for the 3 days preceding the surgery
  Other Names: Magnesium
  Arms: Preoperative oral Magnesium
Drug: Placebo Oral Tablet — Placebo for Magnesium
  Other Names: Placebo
  Arms: Control

SUMMARY:
Post operative atrial fibrillation following coronary surgery (POAF) is a common complication that can affect 10-50% of patients.

Intravenous magnesium, administered per-or post-operatively, reduces the incidence of POAF. However, the effect of preoperative magnesium loading on the incidence of POAF is not yet studied.

200 patients admitted for elective coronary surgery under Cardiopulmonary bypass will be included in this prospective randomized controlled trial.

Treatment group will receive preoperative oral magnesium and control group will receive placebo for 3 days before the planned coronary artery surgery.

The occurrence of POAF will be studied as a main outcome.

DETAILED DESCRIPTION:
Post operative atrial fibrillation following coronary surgery (POAF) is a common complication that can affect 10-50% of patients. It is associated with many complications. POAF increases the postoperative length of stay and increases the cost of hospitalization.

Several studies and meta-analyzes have demonstrated the beneficial effect of intravenous magnesium (Mg), administered per-or post-operatively, in reducing the incidence of POAF. However, the effect of preoperative magnesium loading on the incidence of POAF is not yet studied.

The aim of this study is to study the effect of oral Mg, administered preoperatively, on the incidence of POAF.

Following IRB approval, 200 patients admitted for elective coronary surgery under Cardiopulmonary bypass will be included in this prospective randomized controlled trial. Patients will be allocated inn a 1: 1 ratio in 2 groups:

* Treatment group will receive preoperatively 8 tablets of Mg (3.2 g) per day, at day (-3), day (-2), and day (-1) before the day of planned coronary artery surgery.
* Control group will receive 8 tablets of placebo daily,at day (-3), day (-2), and day (-1) before the day of planned coronary artery surgery.

The anesthetic and surgical management protocols will be identical for both groups. The occurrence of POAF during the 7 postoperative days, the main outcome of the study, will be recorded, including the number of POAF episodes, their duration, recurrence, and the associated ventricular response rate. From a safety point, the occurrence of complications and the length of hospital stay will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Coronary artery disease
* Planned coronary artery surgery
* signed informed consent

Exclusion Criteria:

* Preoperative supraventricular dysrhythmia including atrial fibrillation, either acute or chronic
* Left ventricular EF < 30%
* Urgent surgery
* Redo surgery
* Permanent preoperative pacemaker
* Preoperative anti arrythmia drugs classes I and III
* Post operative inotrope drugs
* Postoperative bradycardia necessitating electrosystolic pacing
* Preoperative heart rate less than 50 bpm
* documented preoperative dysthryroidism
* 2nd and 3rd degree atrioventricular bloc
* Renal failure with GFR < 30 ml/min/1.73 m²

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-11-24 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
postoperative atrial fibrillation | 7 postoperative days
  New onset of atrial fibrillation clinically or telemetry detected and confirmed by EKG

SECONDARY OUTCOMES:
Ventricular response rate | During the atrial fibrillation episodes
  Average ventricular rate during atrial fibrillation episodes
Recurrence of atrial fibrillation | 7 postoperative days
  Relapse of atrial fibrillation following the initial episode

OTHER OUTCOMES:
Length of hospital stay | ranges from 5 to 30 days
  Time from surgery until discharge of the patient
Stroke | 30 postoperative days
  New onset focal neurological deficit following coronary artery surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samia N Madi-Jebara, Principal Investigator — Saint-Joseph University
Locations (1):
- Hotel Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be made available upon request from researchers who need to perform a meta analysis on the subject.
  IPD will be sent directly to the requesting party

REFERENCES:
- [Derived] Tohme J, Sleilaty G, Jabbour K, Gergess A, Hayek G, Jebara V, Madi-Jebara S. Preoperative oral magnesium loading to prevent postoperative atrial fibrillation following coronary surgery: a prospective randomized controlled trial. Eur J Cardiothorac Surg. 2022 Oct 4;62(5):ezac269. doi: 10.1093/ejcts/ezac269. PMID 35451469